CLINICAL TRIAL: NCT02741570
Title: An Open Label, Randomized, Two Arm Phase III Study of Nivolumab in Combination With Ipilimumab Versus Extreme Study Regimen (Cetuximab + Cisplatin/Carboplatin + Fluorouracil) as First Line Therapy in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study of Nivolumab in Combination With Ipilimumab Compared to the Standard of Care (Extreme Regimen) as First Line Treatment in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: CheckMate 651
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-651; 2016-000725-39 (EudraCT Number)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; Ipilimumab; Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab and Ipilimumab (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Extreme Regimen (Active Comparator): Specified dose on specified days
  Interventions: Drug: Cetuximab/Erbitux; Drug: Cisplatin/Platinol; Drug: Carboplatin/Paraplatin; Drug: Fluorouracil/Adrucil

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; Opdivo
  Arms: Nivolumab and Ipilimumab
Biological: Ipilimumab
  Other Names: BMS-734016; Yervoy
  Arms: Nivolumab and Ipilimumab
Drug: Cetuximab/Erbitux
  Arms: Extreme Regimen
Drug: Cisplatin/Platinol
  Arms: Extreme Regimen
Drug: Carboplatin/Paraplatin
  Arms: Extreme Regimen
Drug: Fluorouracil/Adrucil
  Arms: Extreme Regimen

SUMMARY:
The main purpose of this study is to compare nivolumab and ipilimumab with the extreme regimen as first line treatment in patients with recurrent or metastatic squamous cell of the head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent squamous cell carcinoma of the head and neck (oral cavity, oropharynx, hypopharynx & larynx) that is not amenable to curative therapy.
* No prior systemic cancer therapy for recurrent or metastatic disease (except if chemotherapy was part of multimodal treatment completed 6 months prior to enrolment).
* Measurable disease detected by imaging exam (CT or MRI).
* Have tumor tissue for PD L1 expression testing, and for oropharyngeal cancer have results from testing of HPV p16 status.

Exclusion Criteria:

* Metastatic or recurrent carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary, squamous cell carcinoma originating from skin and salivary glands or non squamous histologies (eg. mucosal melanoma).
* No prior treatment with anti PD1, anti PD L1, anti CTLA 4 antibody or any other antibody or drugs targeting T cell costimulation or checkpoint pathways, or cetuximab or EGFR inhibitors in any treatment setting.
* Participants with certain diseases such as active autoimmune disease, type I diabetes, hypothyroidism that needs hormone replacement, active infection, psychiatric disorder.
* Inadequate hematologic, renal or hepatic function.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (133):
- United States (22):
  - Local Institution - 0134, Tucson, Arizona
  - Local Institution - 0135, Duarte, California
  - Local Institution - 0005, Stanford, California
  - Local Institution - 0028, Jacksonville, Florida
  - Local Institution - 0008, Tampa, Florida
  - Local Institution - 0111, Atlanta, Georgia
  - Local Institution - 0006, Chicago, Illinois
  - Local Institution - 0001, Boston, Massachusetts
  - Local Institution - 0080, Boston, Massachusetts
  - Local Institution - 0093, Boston, Massachusetts
  - Local Institution - 0004, Ann Arbor, Michigan
  - Local Institution - 0012, Charlotte, North Carolina
  - Local Institution - 0007, Columbus, Ohio
  - Local Institution - 0010, Langhorne, Pennsylvania
  - Local Institution - 0015, Philadelphia, Pennsylvania
  - Local Institution - 0013, Pittsburgh, Pennsylvania
  - Local Institution - 0139, Dallas, Texas
  - Local Institution - 0009, Houston, Texas
  - Local Institution - 0014, Houston, Texas
  - Local Institution - 0003, Charlottesville, Virginia
  - Local Institution - 0011, Fairfax, Virginia
  - Local Institution - 0125, Morgantown, West Virginia
- Australia (10):
  - Local Institution - 0142, Blacktown, New South Wales
  - Local Institution - 0127, Darlinghurst, New South Wales
  - Local Institution - 0128, Gosford, New South Wales
  - Local Institution - 0019, St Leonards, New South Wales
  - Local Institution - 0077, Brisbane, Queensland
  - Local Institution - 0036, Douglas, Queensland
  - Local Institution - 0021, Elizabeth Vale, South Australia
  - Local Institution - 0022, Clayton, Victoria
  - Local Institution - 0131, Melbourne, Victoria
  - Local Institution - 0020, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0075, Linz
  - Local Institution - 0071, Vienna
- Brazil (8):
  - Local Institution - 0148, Belo Horizonte, Minas Gerais
  - Local Institution - 0121, Ijuí, Rio Grande do Sul
  - Local Institution - 0122, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0120, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0117, Barretos, São Paulo
  - Local Institution - 0123, Sao Jose de Rio Preto, São Paulo
  - Local Institution - 0118, São Paulo
  - Local Institution - 0124, São Paulo
- France (13):
  - Local Institution - 0133, Amiens, Somme
  - Local Institution - 0094, Bordeaux
  - Local Institution - 0140, La Tronche
  - Local Institution - 0090, Lille
  - Local Institution - 0138, Lyon
  - Local Institution - 0054, Lyon
  - Local Institution - 0126, Marseille
  - Local Institution - 0055, Nice
  - Local Institution - 0039, Paris
  - Local Institution - 0088, Paris
  - Local Institution, Paris
  - Local Institution - 0089, Strasbourg
  - Local Institution - 0040, Villejuif
- Germany (10):
  - Local Institution - 0068, Bonn
  - Local Institution - 0078, Freiburg im Breisgau
  - Local Institution - 0067, Hamburg
  - Local Institution - 0092, Hanover
  - Local Institution - 0079, Heidelberg
  - Local Institution - 0074, Leipzig
  - Local Institution - 0070, Mainz
  - Local Institution - 0065, München
  - Local Institution - 0069, Ulm
  - Local Institution - 0066, Würzburg
- Greece (3):
  - Local Institution - 0018, Athens
  - Local Institution - 0017, Nea Kifissia
  - Local Institution - 0051, Thessaloniki
- Local Institution - 0147, Dublin, Dublin, Ireland
- Israel (5):
  - Local Institution - 0062, Haifa
  - Local Institution - 0060, Jerusalem
  - Local Institution - 0063, Petah Tikva
  - Local Institution - 0061, Ramat Gan
  - Local Institution - 0064, Tel Aviv
- Italy (9):
  - Local Institution - 0042, Milan, MI
  - Local Institution - 0043, Torino, TO
  - Local Institution - 0044, Cuneo
  - IRST Meldola, Meldola (FC)
  - Azienda Ospedaliera Universitaria Di Modena, Modena
  - Aorn Dei Colli, Napoli
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliera Di Perugia, Perugia
  - Fondazione Policlinico Universitario A. Gemelli, Roma
- Japan (19):
  - Local Institution - 0106, Nagoya, Aichi-ken
  - Local Institution - 0100, Kashiwa, Chiba
  - Local Institution - 0113, Fukuoka, Fukuoka
  - Local Institution - 0105, Sapporo, Hokkaido
  - Local Institution - 0107, Akashi-shi, Hyōgo
  - Local Institution - 0102, Kobe, Hyōgo
  - Local Institution - 0152, Isehara, Kanagawa
  - Local Institution - 0150, Yokohama, Kanagawa
  - Local Institution - 0151, Natori-shi, Miyagi
  - Local Institution - 0108, Sendai, Miyagi
  - Local Institution - 0146, Osakasayaha, Osaka
  - Local Institution - 0099, Takatsuki-shi, Osaka
  - Local Institution - 0149, Kitaadachi-gun, Saitama
  - Local Institution - 0114, Sunto-gun, Shizuoka
  - Local Institution, Shimotsuke-shi, Tochigi
  - Local Institution - 0153, Bunkyo-ku, Tokyo
  - Local Institution - 0101, Chuo-ku, Tokyo
  - Local Institution - 0104, Koto-ku, Tokyo
  - Local Institution - 0109, Kita-gun
- Mexico (6):
  - Local Institution - 0032, León, Guanajuato
  - Local Institution - 0034, Mexico City, Mexico City
  - Local Institution - 0030, Mexico City, Mexico City
  - Local Institution - 0031, Morelia, Michoacán
  - Local Institution - 0033, Monterrey, Nuevo León
  - Local Institution - 0035, Oaxaca City
- Poland (5):
  - Local Institution - 0037, Bydgoszcz
  - Local Institution - 0023, Gdansk
  - Local Institution - 0129, Gliwice
  - Local Institution - 0026, Krakow
  - Local Institution - 0025, Warsaw
- South Korea (3):
  - Local Institution - 0096, Gangnam-gu
  - Local Institution - 0110, Seoul
  - Local Institution - 0095, Seoul
- Spain (6):
  - Local Institution - 0083, Barcelona
  - Local Institution - 0130, L'Hospitalet Del Llobregat
  - Local Institution - 0085, Madrid
  - Local Institution - 0082, Madrid
  - Local Institution - 0084, Seville
  - Local Institution - 0081, Valencia
- Switzerland (2):
  - Local Institution - 0072, Basel
  - Local Institution - 0073, Zurich
- Taiwan (2):
  - Local Institution - 0097, Taichung
  - Local Institution - 0098, Taipei
- United Kingdom (7):
  - Local Institution - 0049, Newcastle upon Tyne, Durham
  - Local Institution - 0045, London, Greater London
  - Local Institution - 0046, Manchester, Greater Manchester
  - Local Institution - 0047, Southampton, Hampshire
  - Local Institution - 0091, Sutton, Surrey
  - Local Institution - 0050, Birmingham, West Midlands
  - Local Institution - 0132, Sheffield

REFERENCES:
- [Derived] Haddad RI, Harrington K, Tahara M, Ferris RL, Gillison M, Fayette J, Daste A, Koralewski P, Zurawski B, Taberna M, Saba NF, Mak M, Kawecki A, Girotto G, Alvarez Avitia MA, Even C, Toledo JGR, Guminski A, Muller-Richter U, Kiyota N, Roberts M, Khan TA, Miller-Moslin K, Wei L, Argiris A. Nivolumab Plus Ipilimumab Versus EXTREME Regimen as First-Line Treatment for Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck: The Final Results of CheckMate 651. J Clin Oncol. 2023 Apr 20;41(12):2166-2180. doi: 10.1200/JCO.22.00332. Epub 2022 Dec 6. PMID 36473143
- [Derived] Hwang M, Seiwert TY. Are taxanes the future for head and neck cancer? Pragmatism in the immunotherapy era. Lancet Oncol. 2021 Apr;22(4):413-415. doi: 10.1016/S1470-2045(21)00121-2. Epub 2021 Mar 5. No abstract available. PMID 33684371
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 947 participants randomized to receive study treatment. 909 participants received study treatment.
Groups:
- Nivolumab + Ipilimumab: Nivolumab 3 mg/kg IV every 2 weeks + Ipilimumab 1 mg/kg IV every 6 weeks until progression, unacceptable toxicity, or a maximum of 24 months from first nivolumab treatment.
- EXTREME Regimen: Cetuximab 400 mg/m2 IV for the initial dose only, then 250 mg/m2 weekly + cisplatin (100mg/m2) or carboplatin (AUC of 5 mg per milliliter per minute) on Day 1 and fluorouracil (1000 mg/m2 per day for 4 days) every 3 weeks for maximum of 6 cycles followed by maintenance cetuximab at 250 mg/m2 weekly (or every 2 weeks, per local prescribing information) until disease progression or unacceptable toxicity; the choice of cisplatin or carboplatin is at the discretion of the investigator.
Period: Pre-Treatment Period
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Started | 472 | 475
Completed (Continuing into treatment period) | 468 | 441
Not Completed | 4 | 34
Not completed — Other reasons | 0 | 3
Not completed — Participant no longer meets study criteria | 3 | 6
Not completed — Poor/non-compliance | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Participant withdrew consent | 0 | 18
Not completed — Participant request to discontinue study treatment | 0 | 2
Not completed — Adverse event unrelated to study drug | 1 | 0
Not completed — Death | 0 | 1
Not completed — Disease progression | 0 | 1
Period: Treatment Period
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Started | 468 | 441
Completed (Participants continuing in the treatment period) | 0 | 0
Not Completed | 468 | 441
Not completed — Other reasons | 47 | 12
Not completed — Poor/non-compliance | 0 | 2
Not completed — Maximum clinical benefit | 4 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Participant withdrew consent | 9 | 13
Not completed — Participant request to discontinue treatment | 8 | 23
Not completed — Adverse event unrelated to study drug | 41 | 26
Not completed — Death | 9 | 7
Not completed — Study drug toxicity | 55 | 47
Not completed — Disease progression | 294 | 301
Not completed — Administrative reason by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen | Total
Number analyzed (Participants) | 472 | 475 | 947
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (9.7) | 60.9 (9.5) | 60.6 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 310 | 295 | 605
  >= 65 AND < 75 | 134 | 151 | 285
  >= 75 AND < 85 | 26 | 28 | 54
  >= 85 | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 78 | 170
  Male | 380 | 397 | 777
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 43 | 83
  Not Hispanic or Latino | 199 | 207 | 406
  Unknown or Not Reported | 233 | 225 | 458
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 12
  Asian | 58 | 55 | 113
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 7 | 22
  White | 379 | 401 | 780
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Programmed Death-Ligand 1 (PD-L1) With a Combined Positive Score (CPS) ≥20
Description: Overall survival (OS) is defined as the time between randomization and death. For participants without documentation of death, OS will be censored on the last date the participant was known to be alive. Overall survival will be censored at the date of randomization for participants who were randomized but had no follow-up. Survival follow-up will be conducted every 3 months after participants off-treatment date. (Based on Kaplan-Meier estimates)
Time Frame: From randomization to date of death or date the participant was last known to be alive (Up to approximately 55 months)
Population: All randomized PD-L1 CPS >= 20 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 185 | 178
Months | 17.58 [13.77 to 21.98] | 14.59 [12.32 to 15.97]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; p = 0.0469, Log Rank; stratified regular log-rank test; Hazard Ratio (HR) = 0.78, 97.51% CI 2-sided [0.59 to 1.03]

2. Primary Outcome: Overall Survival (OS) in All Randomized Participants
Description: as for outcome 1
Time Frame: From randomization to date of death or date the participant was last known to be alive (Up to approximately 55 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 472 | 475
Months | 13.90 [12.12 to 15.77] | 13.50 [12.55 to 15.21]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; p = 0.4951, Log Rank; stratified regular log-rank test; Cox Proportional Hazard = 0.95, 97.9% CI 2-sided [0.80 to 1.13]

3. Secondary Outcome: Overall Survival (OS) in Randomized Participants With Programmed Death-Ligand 1 (PD-L1) With a Combined Positive Score (CPS) ≥ 1
Description: as for outcome 1
Time Frame: From randomization to date of death or date the participant was last known to be alive (Up to approximately 65 months)
Population: All randomized PD-L1 CPS ≥ 1 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 355 | 372
Months | 15.67 [13.70 to 18.79] | 13.24 [11.07 to 14.59]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; Cox Proportional Hazard = 0.80, 95% CI 2-sided [0.68 to 0.95]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time between the date of randomization and the date of first documented tumor progression, based on Blinded Independent Central Review (BICR) assessments (per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria), or death due to any cause, whichever occurs first. Participants who neither progress nor die will be censored on the date of their last tumor assessment. Participants who receive subsequent anti-cancer therapy prior to documented progression, will be censored on the date of their last tumor assessment prior to subsequent therapy. (Based on Kaplan-Meier Estimates)
  Progression is defined as at least a 20% increase in the sum of diameters of target lesions, in addition the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death (Up to approximately 65 months)
Population: All randomized participants and randomized PD-L1 CPS >= 20 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 472 | 475
Months
  Randomized participants | 3.29 [2.83 to 4.17] | 6.77 [5.78 to 7.00]
  Randomized PD-L1 CPS >= 20 participants: number analyzed (Participants) | 185 | 178
  Randomized PD-L1 CPS >= 20 participants | 5.39 [3.09 to 6.93] | 6.97 [5.78 to 8.67]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; Cox Proportional Hazard = 1.40, 95% CI 2-sided [1.19 to 1.63] — All Randomized Participants
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.77 to 1.30] — All Randomized PD-L1 CPS >= 20 Participants

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria by blinded independent central review (BICR) assessment.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization up to approximately 65 months
Population: All randomized participants and randomized PD-L1 CPS >= 20 participants
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 472 | 475
Percent
  All randomized participants | 24.2 [20.4 to 28.3] | 37.1 [32.7 to 41.6]
  Randomized PD-L1 CPS >= 20 participants: number analyzed (Participants) | 185 | 178
  Randomized PD-L1 CPS >= 20 participants | 34.1 [27.3 to 41.4] | 35.4 [28.4 to 42.9]

6. Secondary Outcome: Duration of Objective Response (DOR)
Description: The time between the first documented response (Complete response (CR) or partial response (PR)) and progression or death, per RECIST 1.1 by blinded independent central review (BICR) assessment. (Based on Kaplan-Meier Estimates)
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to the first documented response (CR or PR) and progression (up to approximately 65 months)
Population: All randomized participants and randomized PD-L1 CPS >= 20 participants with a BOR response of CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 114 | 176
Months
  All randomized participants | 16.59 [9.69 to 29.40] | 5.88 [5.45 to 6.97]
  Randomized PD-L1 CPS >= 20 participants: number analyzed (Participants) | 63 | 63
  Randomized PD-L1 CPS >= 20 participants | 33.51 [12.12 to NA] — Insufficient number of participants with events | 6.97 [5.65 to 10.12]

7. Post Hoc Outcome: Overall Survival (OS) in Participants With Programmed Death-Ligand 1 (PD-L1) With a Combined Positive Score (CPS) ≥20 - Extended Collection
Description: as for outcome 1
Time Frame: From randomization to date of death or date the participant was last known to be alive (Up to approximately 65 months)
Population: All randomized PD-L1 CPS >= 20 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 185 | 178
Months | 17.74 [13.77 to 21.98] | 14.59 [12.32 to 15.97]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.60 to 0.97]

8. Post Hoc Outcome: Overall Survival (OS) in All Randomized Participants - Extended Collection
Description: as for outcome 1
Time Frame: From randomization to date of death or date the participant was last known to be alive (Up to approximately 65 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
Number analyzed (Participants) | 472 | 475
Months | 13.90 [12.12 to 15.77] | 13.50 [12.48 to 15.11]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs EXTREME Regimen; Test type: Superiority; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.82 to 1.08]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from participants first dose to their study completion (up to approximately 65 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 63 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nivolumab + Ipilimumab | EXTREME Regimen
All-Cause Mortality (participants affected / at risk) | 388/472 | 406/475
Serious Adverse Events (participants affected / at risk) | 313/468 | 290/441
Other Adverse Events (participants affected / at risk) | 420/468 | 429/441
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=468) | EXTREME Regimen (N=441)
Anaemia (Blood and lymphatic system disorders) | 1 | 18
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 1
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 24
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 4 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 2 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0
Corneal perforation (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 10 | 2
Constipation (Gastrointestinal disorders) | 2 | 3
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 10
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric haematoma (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 4
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 0
Oral cavity fistula (Gastrointestinal disorders) | 2 | 1
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 6
Subileus (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4
Asthenia (General disorders) | 1 | 3
Chest pain (General disorders) | 1 | 0
Complication associated with device (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 2
Face oedema (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 4 | 6
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 0
Lithiasis (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 7
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2
Pain (General disorders) | 3 | 2
Performance status decreased (General disorders) | 1 | 0
Pneumatosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 9
Stenosis (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 7 | 8
Suprapubic pain (General disorders) | 1 | 0
Swelling face (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 4 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Actinomycosis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 3
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Candida infection (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 4
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 3
Device related sepsis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Emphysematous cystitis (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 2 | 0
Febrile infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 3 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Infective spondylitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 1
Oral infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pleurisy viral (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 25 | 31
Pneumonia aspiration (Infections and infestations) | 8 | 7
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 10 | 10
Septic shock (Infections and infestations) | 3 | 3
Sialoadenitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 3
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vascular access site cellulitis (Infections and infestations) | 0 | 1
Vascular access site infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Device placement issue (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1
Stoma site ulcer (Injury, poisoning and procedural complications) | 0 | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 2
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1
General physical condition abnormal (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 0 | 2
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte depletion (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 5
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 3 | 3
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 101 | 100
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 5
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 3
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 2 | 2
Device occlusion (Product Issues) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Eating disorder (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 7
Anuria (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 3
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 3
Embolism (Vascular disorders) | 1 | 2
Haemorrhage (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 0
Internal haemorrhage (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 2
Vascular rupture (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=468) | EXTREME Regimen (N=441)
Anaemia (Blood and lymphatic system disorders) | 102 | 190
Leukopenia (Blood and lymphatic system disorders) | 6 | 35
Lymphopenia (Blood and lymphatic system disorders) | 17 | 25
Neutropenia (Blood and lymphatic system disorders) | 11 | 131
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 109
Tinnitus (Ear and labyrinth disorders) | 4 | 27
Hyperthyroidism (Endocrine disorders) | 40 | 2
Hypothyroidism (Endocrine disorders) | 86 | 19
Abdominal pain (Gastrointestinal disorders) | 34 | 36
Constipation (Gastrointestinal disorders) | 95 | 157
Diarrhoea (Gastrointestinal disorders) | 104 | 141
Dyspepsia (Gastrointestinal disorders) | 12 | 29
Dysphagia (Gastrointestinal disorders) | 52 | 49
Nausea (Gastrointestinal disorders) | 101 | 226
Stomatitis (Gastrointestinal disorders) | 24 | 104
Vomiting (Gastrointestinal disorders) | 57 | 121
Asthenia (General disorders) | 73 | 106
Fatigue (General disorders) | 123 | 154
Mucosal inflammation (General disorders) | 27 | 137
Oedema peripheral (General disorders) | 30 | 29
Pain (General disorders) | 26 | 15
Pyrexia (General disorders) | 49 | 46
Folliculitis (Infections and infestations) | 6 | 33
Oral candidiasis (Infections and infestations) | 19 | 29
Paronychia (Infections and infestations) | 9 | 95
Pneumonia (Infections and infestations) | 41 | 25
Upper respiratory tract infection (Infections and infestations) | 26 | 19
Alanine aminotransferase increased (Investigations) | 35 | 23
Amylase increased (Investigations) | 32 | 18
Aspartate aminotransferase increased (Investigations) | 39 | 18
Blood alkaline phosphatase increased (Investigations) | 27 | 19
Blood creatinine increased (Investigations) | 17 | 34
Lipase increased (Investigations) | 50 | 19
Neutrophil count decreased (Investigations) | 19 | 66
Platelet count decreased (Investigations) | 7 | 60
Weight decreased (Investigations) | 57 | 81
White blood cell count decreased (Investigations) | 12 | 36
Decreased appetite (Metabolism and nutrition disorders) | 73 | 115
Dehydration (Metabolism and nutrition disorders) | 5 | 26
Hypercalcaemia (Metabolism and nutrition disorders) | 31 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 20
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 45
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 93
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 | 146
Hyponatraemia (Metabolism and nutrition disorders) | 39 | 35
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 21
Neck pain (Musculoskeletal and connective tissue disorders) | 38 | 38
Dizziness (Nervous system disorders) | 20 | 32
Headache (Nervous system disorders) | 30 | 31
Neuropathy peripheral (Nervous system disorders) | 10 | 34
Insomnia (Psychiatric disorders) | 35 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 | 53
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 40
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 23 | 147
Dry skin (Skin and subcutaneous tissue disorders) | 35 | 79
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 38
Rash (Skin and subcutaneous tissue disorders) | 90 | 177
Skin fissures (Skin and subcutaneous tissue disorders) | 4 | 65
Hypotension (Vascular disorders) | 13 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02741570/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02741570/SAP_001.pdf